CLINICAL TRIAL: NCT03667547
Title: An Open-label Single Oral Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of MK-0518 1200 mg (600 mg Tablet × 2) in Healthy Japanese Male Participants
Brief Title: Safety, Tolerability, and Pharmacokinetics of Raltegravir (MK-0518) in Healthy Japanese Male Participants (MK-0518-851)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0518-851; MK-0518-851 (Other: Merck Protocol Number)
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Results first posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Human Immunodeficiency Virus (HIV) Infection
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Raltegravir (Experimental): Participants will receive a single oral dose of raltegravir 1200 mg (600 mg tablet X 2) in a fasted state on Day 0 and will be followed up to 2 weeks
  Interventions: Drug: Raltegravir

INTERVENTIONS:
Drug: Raltegravir — Raltegravir 600 mg tablet
  Other Names: MK-0518; ISENTRESS®

SUMMARY:
This study is designed to evaluate safety, tolerability, and pharmacokinetics of a single 1200-mg dose of raltegravir (MK-0518, ISENTRESS®) in healthy Japanese male participants.

ELIGIBILITY:
Inclusion Criteria:

* Japanese male in good health
* Body mass index (BMI) between 18.5 and 32.0 kg/m^2
* Nonsmoker and has not used nicotine-containing products for over 3 months at the time of screening test.

Exclusion Criteria:

* History of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or neurological (including cerebrovascular stroke and epilepsy) abnormalities or diseases
* Significant emotional problem at the time of screening test or suspected to occur during the conduct of the study, or has a history of clinically significant psychiatric disorder within the last 5 years
* History of malignancy
* History of clinically significant allergies to multiple antigens or severe allergies (e.g., food, drug, and latex [natural rubber] allergies), or has had an anaphylactic reaction or significant intolerability (e.g., systemic allergic reaction) to prescription or non-prescription drugs or food
* Positive for hepatitis B virus surface antigen, hepatitis C virus antibodies, syphilis, or HIV antigen or antibody on the screening test
* Had surgery or donated or lost blood within 4 weeks prior to the screening test
* Participated in another study (clinical trial) within 4 months prior to the screening test
* Consumes greater than 3 glasses of alcoholic beverages (definition of 1 glass: 354 mL for beer, 118 mL for wine, 29.5 mL for distilled spirits) per day
* Consumes greater than 6 servings (definition of 1 serving: equivalent to 120 mg of caffeine) of coffee, tea, cola, energy drinks, or other caffeinated beverages per day
* Regular user of cannabis, any illicit drugs, or has a history of drug or alcohol abuse within 2 years at the time of the screening test. Participants must have a negative predose urine drug screen
* Unable to consent to refrain from the consumption of citrus beverages and foods (e.g., grapefruits) beginning 2 weeks prior to administration of the study drug until the end of post-study examination, and the consumption of all fruit beverages and foods for 24 hours predose and after dosing
* Is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling, or child) who is study site or Sponsor staff directly involved with this study.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2018-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Medical Corporation Houeikai Sekino Clinical Pharmacology Clinic ( Site 0001), Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Raltegravir: Participants received a single oral dose of raltegravir 1200 mg (600 mg tablet X 2) in a fasted state on Day 0 and were followed up to 2 weeks
Period: Overall Study
Arm/Group | Raltegravir
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Raltegravir
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.17 (4.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of a study drug, whether or not considered related to the study drug. The number of participants with an AE was reported.
Time Frame: Up to Day 14 after dosing
Population: All participants who received at least one dose of the study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Raltegravir
Number analyzed (Participants) | 12
Participants | 0

2. Primary Outcome: Number of Participants Discontinued From the Study Due to an AE
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of a study drug, whether or not considered related to the study drug. The number of participants discontinued from the study due to an AE was reported.
Time Frame: Up to Day 14 after dosing
Population: All participants who received at least one dose of the study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Raltegravir
Number analyzed (Participants) | 12
Participants | 0

3. Primary Outcome: Number of Participants With a Serious Adverse Event (SAE)
Description: A SAE is an AE that results in death, is life-threatening, requires or prolongs an existing hospitalization, results in significant disability or incapacity, is a congenital anomaly or birth defect, is another medically important event, is a new cancer, or is an overdose. The number of participants with an SAE was reported.
Time Frame: Up to Day 14 after dosing
Population: All participants who received at least one dose of the study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Raltegravir
Number analyzed (Participants) | 12
Participants | 0

4. Primary Outcome: Number of Participants With a Drug-related AE
Description: The number of participants with a drug-related AE was reported. Causality was be determined by the investigator.
Time Frame: Up to Day 14 after dosing
Population: All participants who received at least one dose of the study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Raltegravir
Number analyzed (Participants) | 12
Participants | 0

5. Secondary Outcome: Area Under the Concentration-Time Curve Up to Infinity (AUC0-∞) of Plasma Raltegravir
Description: Blood samples were collected from pre-dose up to 48 hours post-dose in order to measure the concentration of plasma raltegravir. Values below the lower limit of quantitation were replaced with 0. Area under the concentration-time curve from time zero extrapolated to infinity (AUC0-∞) of plasma raltegravir was calculated based on natural log-transformed values.
Time Frame: Predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, and 48 hours after dosing
Population: Participants meeting the protocol criteria likely to provide data that sufficiently reflects the effect of treatment under the scientific model. These included measures such as the exposure to study drug, the availability of measurements, and the absence of significant protocol deviations.
Measure: Geometric Mean (95% Confidence Interval); unit: (μM•hr)
Arm/Group | Raltegravir
Number analyzed (Participants) | 12
(μM•hr) | 62.8 [41.8 to 94.4]

6. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Raltegravir
Description: Blood samples were collected from pre-dose up to 48 hours post-dose in order to measure the concentration of plasma raltegravir. Values below the lower limit of quantitation were replaced with 0. Maximum plasma concentration (Cmax) of raltegravir was calculated based on natural log-transformed values.
Time Frame: Predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, and 48 hours after dosing
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Arm/Group | Raltegravir
Number analyzed (Participants) | 12
nM | 20163 [12211 to 33291]

7. Secondary Outcome: Plasma Concentration of Raltegravir at 24 Hours After Dosing (C24)
Description: Blood samples were collected at 24 hours post-dose in order to measure the concentration of plasma raltegravir. Values below the lower limit of quantitation were replaced with 0. The plasma concentration of raltegravir at 24 hours after dosing (C24) was calculated based on natural log-transformed values.
Time Frame: 24 hours after dosing
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Arm/Group | Raltegravir
Number analyzed (Participants) | 12
nM | 74.5 [53.9 to 103]

8. Secondary Outcome: Time of Maximum Plasma Concentration (Tmax) of Raltegravir
Description: Blood samples were collected from pre-dose up to 48 hours post-dose in order to measure the concentration of plasma raltegravir. Values below the lower limit of quantitation were replaced with 0. The time at which Cmax of plasma raltegravir is achieved (Tmax) was reported.
Time Frame: Predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, and 48 hours after dosing
Population: as for outcome 5
Measure: Median (Full Range); unit: Hours
Arm/Group | Raltegravir
Number analyzed (Participants) | 12
Hours | 1.75 [0.5 to 4.0]

9. Secondary Outcome: Apparent Plasma Half-life (t1/2) of Raltegravir
Description: Blood samples were collected from pre-dose up to 48 hours post-dose in order to measure the concentration of plasma raltegravir. Values below the lower limit of quantitation were replaced with 0. The apparent plasma half-life (t1/2) of raltegravir was reported.
Time Frame: Predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, and 48 hours after dosing
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Raltegravir
Number analyzed (Participants) | 12
Hours | 7.50 (34.6)

10. Secondary Outcome: Apparent Total Plasma Clearance (CL/F) of Raltegravir
Description: Blood samples were collected from pre-dose up to 48 hours post-dose in order to measure the concentration of plasma raltegravir. Values below the lower limit of quantitation were replaced with 0. The apparent total plasma clearance of raltegravir after oral dosing (CL/F) was reported.
Time Frame: Predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, and 48 hours after dosing
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Raltegravir
Number analyzed (Participants) | 12
L/hr | 39.6 (71.3)

11. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of Raltegravir
Description: Blood samples were collected from pre-dose up to 48 hours post-dose in order to measure the concentration of plasma raltegravir. Values below the lower limit of quantitation were replaced with 0. The apparent volume of distribution of raltegravir during the terminal phase (Vz/F) was reported.
Time Frame: Predose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, and 48 hours after dosing
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Raltegravir
Number analyzed (Participants) | 12
Liters | 429 (81.1)

ADVERSE EVENTS:
Time Frame: Up to 14 days after treatment with study drug
Description: All participants who received at least one dose of the study drug.
Arm/Group | Raltegravir
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, investigators agree to provide all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-10): https://cdn.clinicaltrials.gov/large-docs/47/NCT03667547/Prot_SAP_000.pdf